CLINICAL TRIAL: NCT05567822
Title: The Effect of Intraoperative Esmolol Administration on Postoperative Recovery and Chronic Pain
Brief Title: The Impact of Esmolol Administration on Postoperative Recovery
Acronym: esmolol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Professor of Anesthesiology, Aretaieion University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 89/24-03-2022
Record Dates: First submitted 2022-10-01; First posted 2022-10-05 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Pain, Acute; Pain, Postoperative; Pain, Chronic Post-Surgical; Esmolol; Inguinal Hernia Repair; Analgesia; Nociceptive Pain
MeSH Terms: conditions — Acute Pain; Pain, Postoperative; Agnosia; Nociceptive Pain | interventions — esmolol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- esmolol group (Active Comparator): loading dose of esmolol 0.05 mL/kg and maintenance dose of esmolol 0.3 mL/kg/h
  Interventions: Drug: Esmolol Hydrochloride
- placebo group (Placebo Comparator): loading dose of 0.9% sodium chloride 0.05 mL/kg and maintenance dose of 0.9% sodium chloride 0.3 mL/kg/h
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Esmolol Hydrochloride — In the esmolol group, patients will receive a bolus dose of esmolol followed by a continuous infusion of esmolol intraoperatively
  Arms: esmolol group
Drug: normal saline — In the placebo group, patients will receive a bolus dose of normal saline followed by a continuous infusion of normal saline intraoperatively
  Arms: placebo group

SUMMARY:
The aim of this study will be to investigate the effect of a continuous infusion of low dose esmolol on intraoperative and postoperative opioid consumption, as well as on postoperative recovery and chronic pain

DETAILED DESCRIPTION:
Contemporary anaesthesiology requires the quest of ways to restrict the use of opioids, which aim at the alleviation of severe postoperative and chronic pain. This is not only due to the side effects involved but also to the epidemic dimensions their use entails. Esmolol, an extremely short-acting cardioselective antagonist of β1 adrenergic receptors, is effectively used in order to attenuate the stress response and minimize undesirable perioperative hemodynamic changes. More specifically, esmolol has been used effectively to reduce pain during induction of anesthesia with propofol and treat tachycardia and hypertension during laryngoscopy. However, recent studies also highlight a possible antinociceptive and/or analgesic effect of esmolol. Therefore, The aim of this study will be to investigate the effect of a continuous infusion of low dose esmolol on intraoperative and postoperative opioid consumption, as well as on postoperative recovery and chronic pain

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* American Society of Anesthesiologists (ASA) classification I-II
* elective inguinal hernia repair

Exclusion Criteria:

* body mass index (BMI) >35 kg/m2
* β-blocker administration preoperatively
* systematic use of analgesic agents preoperatively
* chronic pain syndromes preoperatively
* neurological or psychiatric disease on treatment
* pregnancy
* severe hepatic or renal disease
* history of cardiovascular diseases/ arrhythmias/ conduction abnormalities
* hemodynamic instability
* drug or alcohol abuse
* language or communication barriers
* lack of informed consent
* bilateral inguinal hernia repair

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
pain score 3 hours postoperatively | 3 hours postoperatively
  pain score by the use of Numeric Rating Scale (NRS) 3 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 6 hours postoperatively | 6 hours postoperatively
  pain score by the use of Numeric Rating Scale (NRS) 6 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 24 hours postoperatively | 24 hours postoperatively
  pain score by the use of Numeric Rating Scale (NRS) 24 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"

OTHER OUTCOMES:
pain score on arrival to Post-Anesthesia Care Unit (PACU) | immediately postoperatively
  pain score by the use of Numeric Rating Scale (NRS) on arrival to PACU, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score at discharge from Post-Anesthesia Care Unit (PACU) | at discharge from Post Anesthesia Care Unit (PACU), approximately 1 hour postoperatively]
  pain score by the use of Numeric Rating Scale (NRS) at discharge from PACU, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
sevoflurane consumption during general anesthesia | change of sevoflurane vaporizer weight from before induction to end of anesthesia, an average period of 1-2 hours
  the sevoflurane vaporizer will be weighed before anesthetic induction and at the end of anesthesia and consequently sevoflurane consumption during anesthesia will be determined
time to first request for analgesia | during stay in Post-Anesthesia Care Unit (PACU), approximately 1 hour postoperatively
  the time for the first patient request for analgesia will be noted
morphine consumption in Post-Anesthesia Care Unit (PACU) | immediately postoperatively
  mg of morphine requested during patient PACU stay
tramadol consumption in the first 24 hours | 24 hours postoperatively
  patients will be followed for cumulative tramadol consumption for 24 hours postoperatively
fentanyl requirement during surgery | intraoperatively
  dose of required fentanyl intraoperatively to maintain systolic arterial blood pressure and heart rate within the 20% of baseline value
time to emergence | up to 2 hours after start of surgery
  time from sevoflurane discontinuation to first patient response (eye opening)
time to extubation | up to 2 hours after start of surgery
  time from sevoflurane discontinuation to tracheal extubation
Post Anesthesia Care Unit (PACU) duration of stay | immediately postoperatively
  duration of patient stay at PACU
sedation on arrival to Post-Anesthesia Care Unit | immediately postoperatively
  sedation will be assessed with a 5-point sedation scale, where: 1, patient perfectly conscious; 2, patient feels a little drowsy; 3, patient seems to be sleeping but immediately reacts to verbal stimulation; 4, patient seems to be sleeping but slowly reacts to verbal stimulation and 5, patient seems to be sleeping and does not react to verbal stimulation but does react to a stimulus such as shaking or pain
sedation at discharge from Post-Anesthesia Care (PACU) Unit | at discharge from Post Anesthesia Care Unit (PACU), approximately 1 hour postoperatively
  sedation will be assessed with a 5-point sedation scale, where: 1, patient perfectly conscious; 2, patient feels a little drowsy; 3, patient seems to be sleeping but immediately reacts to verbal stimulation; 4, patient seems to be sleeping but slowly reacts to verbal stimulation and 5, patient seems to be sleeping and does not react to verbal stimulation but does react to a stimulus such as shaking or pain
side effects postoperatively | 48 hours postoperatively
  patients will be monitored for side-effects of the administered agents postoperatively
satisfaction from analgesia | at discharge from Post Anesthesia Care Unit, approximately 1 hour postoperatively
  satisfaction from postoperative analgesia on a four-point Likert scale with 1 marked as minimal satisfaction and 4 as maximal satisfaction
change from baseline in Quality of Recovery (QoR)-15 score after surgery | 24 hours postoperatively
  The QoR-15 is a quality of recovery scale that consists of 15 questions (items),including questions regarding pain (2 items), physical comfort (5 items), self-care ability (2 items), psychological support (2 items) and emotional state (4 items). Every item is scored on a scale of 10, with the lowest total score of 0 and the highest score of 150. The higher the score, the better the recovery quality of the patient
sleep quality | 24 hours postoperatively
  subjective evaluation of sleep quality by patients, based on a sleep questionnaire (evaluation of sleep duration, number of nocturnal awakenings and marking of sleep quality)
first mobilization after surgery | 24 hours postoperatively
  patients will be questioned regarding the time at which they mobilized after surgery
gastrointestinal recovery after surgery | 24 hours postoperatively
  patients will be questioned regarding the time they first felt enteral sounds and the time they had their first flatus after surgery
first fluid intake | 24 hours postoperatively
  patients will be questioned regarding the time they had their first fluid intake
first solid intake | 24 hours postoperatively
  patients will be questioned regarding the time they had their first solid intake
hospitalization time | 96 hours postoperatively
  duration of hospital stay after surgery in hours
incidence of chronic pain 1 month after surgery | 1 month after surgery
  occurrence of chronic pain at the site of the operation 1 month after surgery, with the use of the Numeric Rating Scale (NRS), at rest and during movement
incidence of chronic pain 3 months after surgery | 3 months after surgery
  occurrence of chronic pain at the site of the operation 3 months after surgery, with the use of the Numeric Rating Scale (NRS), at rest and during movement
duration of nociception level<25 intraoperatively | intraoperatively
  nociception level (NOL) is a device that measures the status of analgesia intraoperatively. Levels<25 suggest adequate intraoperatively analgesia
change from baseline in cortisol levels after surgery | during patient stay in the Post Anesthesia Care Unit, approximately 2 hours postoperatively
  blood samples will be collected to measure the variation in cortisol levels from the induction of anesthesia till the arrival of the patient to the Post Anesthesia CAre Unit
change from baseline in prolactin levels after surgery | during patient stay in the Post Anesthesia Care Unit, approximately 2 hours postoperatively
  blood samples will be collected to measure the variation in prolactin levels from the induction of anesthesia till the arrival of the patient to the Post Anesthesia CAre Unit
change from baseline in lactate levels after surgery | during patient stay in the Post Anesthesia Care Unit, approximately 2 hours postoperatively
  blood samples will be collected to measure the variation in lactate levels from the induction of anesthesia till the arrival of the patient to the Post Anesthesia CAre Unit

CONTACTS AND LOCATIONS:
Locations (1):
- Evangelismos General Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Egan TD. Are opioids indispensable for general anaesthesia? Br J Anaesth. 2019 Jun;122(6):e127-e135. doi: 10.1016/j.bja.2019.02.018. Epub 2019 Mar 28. PMID 31104756
- [Background] Salome A, Harkouk H, Fletcher D, Martinez V. Opioid-Free Anesthesia Benefit-Risk Balance: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Clin Med. 2021 May 12;10(10):2069. doi: 10.3390/jcm10102069. PMID 34065937
- [Background] Bahr MP, Williams BA. Esmolol, Antinociception, and Its Potential Opioid-Sparing Role in Routine Anesthesia Care. Reg Anesth Pain Med. 2018 Nov;43(8):815-818. doi: 10.1097/AAP.0000000000000873. PMID 30216240
- [Background] Gelineau AM, King MR, Ladha KS, Burns SM, Houle T, Anderson TA. Intraoperative Esmolol as an Adjunct for Perioperative Opioid and Postoperative Pain Reduction: A Systematic Review, Meta-analysis, and Meta-regression. Anesth Analg. 2018 Mar;126(3):1035-1049. doi: 10.1213/ANE.0000000000002469. PMID 29028742
- [Background] Watts R, Thiruvenkatarajan V, Calvert M, Newcombe G, van Wijk RM. The effect of perioperative esmolol on early postoperative pain: A systematic review and meta-analysis. J Anaesthesiol Clin Pharmacol. 2017 Jan-Mar;33(1):28-39. doi: 10.4103/0970-9185.202182. PMID 28413270
- [Background] Andresen K, Rosenberg J. Management of chronic pain after hernia repair. J Pain Res. 2018 Apr 5;11:675-681. doi: 10.2147/JPR.S127820. eCollection 2018. PMID 29670394